CLINICAL TRIAL: NCT04876040
Title: A Multi-Center Randomized-Controlled Trial To Evaluate The Safety And Feasibility of The Delivery Of Intracoronary Hyperoxemic Supersaturated Oxygen Therapy For 60 Minutes In Patients With St Elevation Myocardial Infarction (STEMI) And Cardiogenic Shock After Successful Reperfusion (Via PCI) ≤ Six Hours After Symptom Onset Compared To Standard Therapy
Brief Title: Incorporating Supersaturated Oxygen in Shock
Acronym: ISO-SHOCK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: TherOx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISO-SHOCK
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cardiogenic Shock; STEMI
Keywords: Supersaturated Oxygen; SSO2
MeSH Terms: conditions — Shock, Cardiogenic; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PCI+Impella plus SSO2 (Experimental): Patients who present with STEMI-CS will undergo treatment with Impella, followed by PCI. Subjects are then immediately treated post-procedure with an infusion of SSO2 Therapy for a duration of 60 minutes.
  Interventions: Device: SSO2 Downstream System; Procedure: PCI + Impella
- PCI+Impella (Active Comparator): Patients who present with STEMI-CS will undergo treatment with Impella, followed by PCI. Subjects are then immediately treated with Standard of Care.
  Interventions: Procedure: PCI + Impella

INTERVENTIONS:
Device: SSO2 Downstream System — 60-min adjunctive reperfusion of hyperoxemic blood into target coronary artery, immediately following revascularization by means of PCI with stenting.
  Arms: PCI+Impella plus SSO2
Procedure: PCI + Impella — Standard of Care Intervention

SUMMARY:
A multi-center, prospective randomized (1:1) pilot and feasibility study to evaluate the safety and feasibility of supersaturated oxygen (SSO2) therapy delivered for 60 minutes selectively into the culprit coronary artery of patients presenting with ST elevation myocardial infarction and cardiogenic shock (STEMI-CS) treated using a shock protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet ALL of the following criteria:

GENERAL INCLUSION CRITERIA: Candidates for this study must meet ALL of the following criteria prior to randomization:

Pre-PCI:

1. The patient must be ≥18 years of age.
2. Symptoms of acute myocardial infarction (AMI) with ECG and/or biomarker evidence of ST-segment elevation myocardial infarction (STEMI).
3. Cardiogenic shock is defined by the presence of at least 2 of the below criteria:

   * Hypotension due to a primary cardiac cause (systolic blood pressure [SBP] <90 mmHg refractory to urgent medical care and/or not responsive to initial medical care or requiring inotropes or vasopressors or mechanical circulatory support to maintain SBP >90 mmHg)
   * Signs of end organ hypoperfusion (cool extremities, oliguria or anuria, or elevated lactate levels)
   * Hemodynamic criteria represented by cardiac index <2.2 L/min/m2 or cardiac power output (CPO) <0.6 W.
4. Patient had pulmonary artery catheters placed for hemodynamic monitoring for clinical reasons
5. Patient is treated with mechanical circulatory support with an Impella CP.
6. Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided and signed written or remote/electronic informed consent, approved by the appropriate Institutional Review Board (IRB).
7. Patient or legally authorized representative and his/her physician agree to all required follow-up procedures and visits.

   ANGIOGRAPHIC INCLUSION CRITERIA: These are evaluated after the patient has undergone cardiac catheterization and PCI and has provided signed Informed Consent:
8. Based on coronary anatomy, PCI is indicated for revascularization of the culprit lesion(s) with use of a commercially available coronary stent (bare metal or drug-eluting, at operator discretion).
9. Successful angioplasty with stenting is completed <6 hrs from AMI symptom onset, as documented by less than 30% diameter residual angiographic stenosis within all treated culprit lesions with TIMI 2 or 3 flow and no major complications such as perforation.
10. For coronary intervention, intravenous antiplatelet agents were used
11. Expected ability to place the SSO2 delivery catheter in the coronary ostium to deliver SSO2 Therapy with stable, coaxial alignment.
12. Systemic arterial pO2 greater than or equal to 80 mmHg as measured by arterial blood gas (may be repeated if low after supplemental O2 administration).

Exclusion Criteria:

* Patients will be excluded if ANY of the following conditions apply:

GENERAL EXCLUSION CRITERIA

Pre-PCI:

1. A surgical procedure is planned during the first 30 days post-enrollment.
2. Contraindication to MRI imaging, including any of the following:

   1. Non-MRI compatible cardiac pacemaker or implantable defibrillator;
   2. Non-MRI compatible aneurysm clip or other metallic implants;
   3. Neural Stimulator (i.e., TENS unit);
   4. Any implanted or magnetically activated device (insulin pump);
   5. Any type of non-MRI compatible ear implant;
   6. Metal shavings in the orbits;
   7. Any indwelling metallic foreign body, shrapnel, or bullet;
   8. Any condition contraindicating MRI, including claustrophobia;
   9. Inability to follow breath hold instructions or to maintain a breath hold for >15 seconds; and
   10. Known hypersensitivity or contraindication to gadolinium contrast.
3. All unwitnessed out of hospital cardiac arrest or any witnessed cardiac arrest in which return of spontaneous circulation (ROSC) is not achieved within 30 minutes or any neurological injury
4. Evidence of anoxic brain injury on admission (including posturing, seizures, loss of brain stem reflexes)
5. Use of IABP
6. Septic, anaphylactic, hemorrhagic, or neurologic causes of shock
7. Non-ischemic causes of shock/hypotension (pulmonary embolism, pneumothorax, myocarditis, tamponade, etc.)
8. Known previous myocardial infarction, in the same territory as present AMI
9. Active bleeding for which mechanical circulatory support is contraindicated.
10. Patient has history of bleeding diathesis or coagulopathy (including heparin induced thrombocytopenia), or refusal to receive blood transfusions if necessary.
11. Contraindication to intravenous systemic anticoagulation
12. Mechanical complications of AMI (acute ventricular septal defect (VSD) or acute papillary muscle rupture)
13. Known left ventricular thrombus for which mechanical circulatory support with Impella is contraindicated
14. Mechanical aortic prosthetic valve or self-expanding TAVR (note: prior bioprosthetic surgical valve or balloon-expandable TAVR implanted >24 hours pre-procedure is acceptable)
15. Known impaired renal function (creatinine clearance <30 ml/min/1.73 m2 by the MDRD formula) or on dialysis.
16. History of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke.
17. Stroke or transient ischemic attack within the past six (6) months, or any permanent neurological defect.
18. Gastrointestinal or genitourinary bleeding within the last two (2) months.
19. Any major surgery (including CABG) within six weeks of enrollment.
20. Patient has received any organ transplant or is on a waiting list for any organ transplant.
21. Patient has other medical illness (e.g., cancer, dementia) with life expectancy of less than one year.
22. Patient has a known hypersensitivity or contraindication to any of the required study medications or contrast that cannot be adequately premedicated.
23. Patient with severe peripheral arterial disease in whom mechanical circulatory support cannot be safely established (or who require a smaller device such as an IABP).
24. Severe known cardiac valvular stenosis or insufficiency, pericardial disease, or cardiomyopathy.
25. Patient is a member of a vulnerable population or has any significant medical or social condition which in the investigator's opinion may interfere with the patient's participation in the study or ability to comply with follow-up procedures, including MRI (e.g. alcoholism, dementia, lives far from the research center, etc.).
26. Current participation in other investigational device or drug study that has not reached its primary endpoint.
27. Symptoms consistent with isolated right ventricular cardiogenic shock (this study is intended to enroll patients experiencing cardiogenic shock from predominant left ventricular dysfunction).
28. Previous enrollment in this study.
29. Subject is currently hospitalized for definite or suspected COVID-19.

    ANGIOGRAPHIC EXCLUSION CRITERIA: These are evaluated after the patient has provided signed Informed Consent and has undergone cardiac catheterization and PCI if indicated:
30. Left ventriculography or high-quality echocardiography (at least one of which is mandatory either before or after PCI, but in all cases before randomization) demonstrates severe mitral regurgitation with concerns of papillary muscle rupture, a ventricular septal defect, a pseudoaneurysm, aortic dissection or other mechanical complications of MI.
31. Any unrevascularized left main or ostial right coronary artery stenosis >50%, which would preclude use of the delivery catheter.
32. Presence of a non-stented coronary dissection with NHLBI grade >B upon completion of the PCI procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
All cause mortality at 30-days in the SSO2 group rate compared with the control group rate | 30 days
  Primary Safety Endpoint

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Baptist Health South Florida, Miami, Florida
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - WakeMed, Raleigh, North Carolina
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No